CLINICAL TRIAL: NCT01989000
Title: The Role of the Tumor Microenvironment of Pancreatic Cancer to Predict Treatment Outcome
Acronym: MIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, M.D., Ph.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL45913.018.13
Record Dates: First submitted 2013-11-08; First posted 2013-11-20 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Hypoxia; Vasculature; Stroma
MeSH Terms: conditions — Pancreatic Neoplasms; Hypoxia | interventions — gadobutrol; 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol; Gemcitabine; Radiotherapy; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant radiochemotherapy (Active Comparator): Patients elected for neoadjuvant radiochemotherapy undergo DWI-MRI, DCE-MRI (Gadobutrol),T2*-MRI and [F-18]HX4 PET/CT imaging within two weeks before start of the chemoradiation and again after radiochemotherapy (Gemcitabine/Radiotherapy), within two weeks before surgery (Pancreaticoduodenectomy).
  Interventions: Drug: Gadobutrol; Drug: [F-18]HX4; Drug: Gemcitabine; Radiation: Radiotherapy; Procedure: Pancreaticoduodenectomy
- Primary Surgery (Active Comparator): Patients elected for primary surgery undergo DWI-MRI, DCE-MRI (Gadobutrol),T2*-MRI and [F-18]HX4 PET/CT imaging within two weeks before surgery (Pancreaticoduodenectomy).
  Interventions: Drug: Gadobutrol; Drug: [F-18]HX4; Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Drug: Gadobutrol — 0.1 ml/kg Gadovist is administered at 5 ml/s followed by a 15 ml saline flush
  Other Names: Gadovist
Drug: [F-18]HX4 — 400 MBq [F-18]HX4, is administered in a single intravenous bolus injection, followed by a saline flush.
  Other Names: [18 F]-3-Fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-; 1H-1,2,3-triazol-1-yl)propan-1-ol
Drug: Gemcitabine — 1000 mg/m2/dose on day 1 and 8 in 2 cycles of 21 days (three weeks) each, one cycle before and one cycle after radiochemotherapy. During radiotherapy gemcitabine is administered at 1000 mg/m2/dose on day 1, 8 and 15.
  Other Names: Gemzar
  Arms: Neoadjuvant radiochemotherapy
Radiation: Radiotherapy — A hypofractionated scheme of 15 fractions of 2.4 Gy in three weeks will be applied, combined with the second course of gemcitabine.
  Arms: Neoadjuvant radiochemotherapy
Procedure: Pancreaticoduodenectomy
  Other Names: PPPD; Whiple

SUMMARY:
Pancreatic cancer is a highly lethal disease. Patients with resectable or borderline resectable disease may benefit from preoperative radiochemotherapy. However, only a subset of patients will respond to this potentially toxic and expensive treatment. Therefore, novel predictive markers are needed to determine treatment efficacy at an early stage. Preferably, these markers could be determined non-invasively and provide insight into the biology of pancreatic cancer. Pancreatic cancers are heterogeneous tumors. The tumor microenvironment is often characterized by large amounts of stroma, hypovascularization, and hypoxia. As these three factors can all contribute to treatment resistance, a quantitative assessment of these markers may aid in the prediction of response to preoperative radiochemotherapy. Moreover, these assessments may have prognostic value. Finally, further insight into the interrelation of these aspects of the tumor microenvironment can contribute to the evaluation of new targeted treatment options. Tumor cellularity and extracellular matrix composition can be assessed non-invasively in vivo by diffusion weighted magnetic resonance imaging (DWI) and tumor vascularity can be assessed by dynamic contrast enhanced magnetic resonance imaging (DCE-MRI). Finally, tumor hypoxia can be evaluated by T2* MRI and PET-CT, using the 18F-labeled hypoxic marker HX4.

Objective of the study:

The primary aim of the study is to assess whether DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT predict overall survival in patients with pancreatic cancer treated with surgery and adjuvant chemotherapy or with neoadjuvant radiochemotherapy, surgery and adjuvant chemotherapy. Secondary aims of the study include the assessment of the predictive value of DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT for pathological response to neoadjuvant chemoradiation, the correlation of DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT with histopathological assessment of tumor stroma, vascularization, and hypoxia, and the assessment of the predictive value of these histopathological markers for overall survival.

DETAILED DESCRIPTION:
Background of the study:

Pancreatic cancer is a highly lethal disease. Patients with resectable or borderline resectable disease may benefit from preoperative radiochemotherapy. However, only a subset of patients will respond to this potentially toxic and expensive treatment. Therefore, novel predictive markers are needed to determine treatment efficacy at an early stage. Preferably, these markers could be determined non-invasively and provide insight into the biology of pancreatic cancer. Pancreatic cancers are heterogeneous tumors. The tumor microenvironment is often characterized by large amounts of stroma, hypovascularization, and hypoxia. As these three factors can all contribute to treatment resistance, a quantitative assessment of these markers may aid in the prediction of response to preoperative radiochemotherapy. Moreover, these assessments may have prognostic value. Finally, further insight into the interrelation of these aspects of the tumor microenvironment can contribute to the evaluation of new targeted treatment options. Tumor cellularity and extracellular matrix composition can be assessed non-invasively in vivo by diffusion weighted magnetic resonance imaging (DWI) and tumor vascularity can be assessed by dynamic contrast enhanced magnetic resonance imaging (DCE-MRI). Finally, tumor hypoxia can be evaluated by T2* MRI and PET-CT, using the 18F-labeled hypoxic marker HX4.

Objective of the study:

The primary aim of the study is to assess whether DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT predict overall survival in patients with pancreatic cancer treated with surgery and adjuvant chemotherapy or with neoadjuvant radiochemotherapy, surgery and adjuvant chemotherapy. Secondary aims of the study include the assessment of the predictive value of DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT for pathological response to neoadjuvant chemoradiation, the correlation of DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT with histopathological assessment of tumor stroma, vascularization, and hypoxia, and the assessment of the predictive value of these histopathological markers for overall survival.

Study design:

The target population will be recruited from the the Academic Medical Centre (AMC) and Erasmus MC. First, to assess reproducibility, patients with pancreatic cancer will undergo MRI twice, once in the AMC and once in the EMC. Next, 40 consecutive patients that will undergo surgery+adjuvant treatment will have MRI and 18F-HX4-PET/CT measurements once to assess the value of the techniques to predict outcome of standard treatment. 40 patients who will undergo preoperative radiochemotherapy will have MRI and 18F-HX4-PET/CT at baseline, and 1 week before surgery. We will assess the relative contribution of each imaging method as well as the integrated use of these methods as predictive markers for survival and pathological response to treatment. Tumor tissue from resected patients will be analyzed for markers of tumor vascularization (CD31, VEGF), hypoxia (HIF1alfa, GLUT1, CA9), and stromal activation (smooth muscle actin, markers for Hedgehog pathway activity). Results will be correlated with imaging parameters, as well as patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic tumors, with histological or cytological proof of adenocarcinoma or a high suspicion on CT imaging.
* Tumor size ≥ 1cm.
* WHO-performance score 0-2.
* Scheduled for surgery or neo-adjuvant chemotherapy/radiation followed by surgery. For the reproducibility part of the study, patients who will not undergo surgery, may be included, too.
* Written informed consent.

Exclusion Criteria:

* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol.
* Contra-indications for MR scanning, including patients with a pacemaker, cochlear implant or neurostimulator; patients with non-MR compatible metallic implants in their eye, spine, thorax or abdomen; or a non-MR compatible aneurysm clip in their brain; patients with severe claustrophobia.
* Renal failure (GFR < 30 ml/min) hampering safe administration of Gadolinium containing MR contrast agent.
* For the reproducibility part of the protocol: surgery, radiation and/or chemotherapy foreseen within the timeframe needed for MR scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of pretreatment DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT on overall survival in patients with pancreatic cancer treated with surgery and adjuvant chemotherapy or with neoadjuvant radiochemotherapy, surgery and adjuvant chemotherapy. | Within two weeks before start radiochemotherapy or within two weeks before surgery
  DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor. 18F-HX4-PET/CT: SUVmean of the whole tumor.

SECONDARY OUTCOMES:
Predictive value of pretreatment DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT on recurrence free survival in patients with pancreatic cancer treated with surgery and adjuvant chemotherapy or with neoadjuvant radiochemotherapy, surgery and adjuvant chemotherapy. | Within two weeks before start radiochemotherapy or within two weeks before surgery
  DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor. 18F-HX4-PET/CT: SUVmean of the whole tumor.
Predictive value of pretreatment DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT on pathological response in patients with pancreatic cancer treated with neoadjuvant radiochemotherapy | Within two weeks before start radiochemotherapy
  DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor. 18F-HX4-PET/CT: SUVmean of the whole tumor.
Predictive value of changes in DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT parameters after radiochemotherapy on pathological response in patients with pancreatic cancer treated with neoadjuvant radiochemotherapy | Within two weeks before start radiochemotherapy and within two weeks before surgery
  DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor. 18F-HX4-PET/CT: SUVmean of the whole tumor.
Predictive value of changes in DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT parameters after radiochemotherapy on recurrence-free survival in patients with pancreatic cancer treated with neoadjuvant radiochemotherapy, surgery and adjuvant chemotherapy | Within two weeks before start radiochemotherapy and within two weeks before surgery
  DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor. 18F-HX4-PET/CT: SUVmean of the whole tumor.
Immunohistochemically determined parameters of the tumor microenvironment assessed after resection of the pancreatic tumor to predict overall and recurrence-free survival | Within 1h after surgery
  Tumor stroma: SMA (DAKO M0851, 1:800); collagen (picro-sirius red), SHH (H160 anti-SHH, 1:500).
  Tumor angiogenesis: VEGF (VEGF RB-9031, 1:200) and CD34 (Immunotech 0787, 1:600).
  Tumor hypoxia: HIF-1α (Abcam 2185, 1:750), GLUT1 (NeoMarkers RB-90522,1:500), and CA-IX (Mo-anti-CA-IX m75, 1:25).
  Measure: Percentage of staining of the total tumor area
Immunohistochemically determined parameters of the tumor microenvironment assessed in a pretreatment tumor biopsy to predict overall and recurrence-free survival | Within 1h after surgery
  Tumor stroma: SMA (DAKO M0851, 1:800); collagen (picro-sirius red), SHH (H160 anti-SHH, 1:500).
  Tumor angiogenesis: VEGF (VEGF RB-9031, 1:200) and CD34 (Immunotech 0787, 1:600).
  Tumor hypoxia: HIF-1α (Abcam 2185, 1:750), GLUT1 (NeoMarkers RB-90522,1:500), and CA-IX (Mo-anti-CA-IX m75, 1:25).

OTHER OUTCOMES:
DWI, DCE-MRI, T2*, and 18F-HX4-PET/CT parameters obtained just before surgery correlate with immunohistochemically determined parameters of the tumor microenvironment assessed in tumor tissue obtained at surgery | Within two week before surgery and within 1h after surgery
  See before
Immunohistochemically determined parameters of the tumor microenvironment assessed in pretreatment tumor biopsies and post-surgery resection material correlate | Within 4 weeks before start treatment and within 1h after surgery
  See before

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland